CLINICAL TRIAL: NCT00977860
Title: Prospective Evaluation Of Hypofractionated Stereotactic Body Radiotherapy For Low And Intermediate Risk Prostate Cancer
Brief Title: Hypofractionated SBRT For Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Olson (Other)
Responsible Party: Sponsor-Investigator, Adam Olson, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 09-031
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; Stereotactic; Radiosurgery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SBRT (Other)
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — 36.25 Gy in 5 fractions (7.25 Gy/fx) delivered over a 2-week period
  Other Names: CyberKnife; Trilogy; True Beam; Radiosurgery

SUMMARY:
The purpose of this study is to determine, in both low-risk and intermediate-risk cohorts, the rates of acute and late grade 3 or higher gastrointestinal and genitourinary toxicity observed during a 24 month follow up and to estimate the rate of biochemical Disease-Free Survival, Phoenix and American Society for Therapeutic Radiology and Oncology definitions, at 2 years following hypofractionated stereotactic body radiation therapy for low and intermediate risk prostate cancer.

DETAILED DESCRIPTION:
Radiosurgery should be ideal for treating prostate cancer because:

* targeting accuracy for static targets is excellent, with an error of about 1mm,
* it can adjust for intra-fractional organ motion, reducing the volume of the target PTV and therefore the dose to surrounding organs,
* by using over one-hundred non-conplanar beams, the dose gradient between the prostate and surrounding tissues may be superior to that achieved with conventional linear accelerators,
* the radiobiology of prostate cancer may favor large dose per fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma
* Gleason score 2-7
* Biopsy within one year of date of registration
* Clinical stage T1b-T2b, N0-Nx, M0-Mx (AJCC 6th Edition)
* T-stage and N-stage determined by physical exam and available imaging studies (ultrasound, CT, and/or MRI)
* M-stage determined by physical exam, CT or MRI. Bone scan not required unless clinical findings suggest possible osseous metastases.
* PSA ≤ 20 ng/dL
* Patients belonging in one of the following risk groups:
* Low: CS T1b-T2a and Gleason 2-6 and PSA ≤ 10, or
* Intermediate: CS T2b and Gleason 2-6 and PSA ≤ 10, or CS T1b-T2b, and Gleason 2-6 and PSA ≤ 20 ng/dL, or Gleason 7 and PSA ≤ 10 ng/dL
* Prostate volume: ≤ 100 cc
* Determined using: volume = π/6 x length x height x width
* Measurement from CT or ultrasound ≤90 days prior to registration.
* ECOG performance status 0-1
* Completion of patient questionnaires:FACT-G questionnaire, AUA questionnaire, EPIC-26 questionnaire, SHIM questionnaire, Utilization of Sexual Medications/Devices questionnaire
* Consent signed.

Exclusion Criteria:

* Prior prostatectomy or cryotherapy of the prostate
* Prior radiotherapy to the prostate or lower pelvis
* Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.
* Chemotherapy for a malignancy in the last 5 years.
* History of an invasive malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years.
* Hormone ablation for two months prior to enrollment, or during treat

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Olson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Hillman Cancer Center - Shadyside Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBRT
Started | 163
Completed | 163
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SBRT
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.80 (6.929)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 162
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 148
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Grade 3 or Higher GI and GU Toxicities
Description: Number of patients experiencing acute grade 3 or higher GI and GU toxicities. Acute toxicities are those occurring within 90 days of start of treatment, assessed using the NCI Common Toxicity Criteria (CTCAE) version 3.0.
Time Frame: Up to 90 days
Population: Patients that received SBRT therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Rate of Late Grade 3 or Higher GI and GU Toxicities
Description: Number of patients experiencing late grade 3 or higher GI and GU toxicities. Late toxicities are those occurring after 90 days post start of treatment, assessed using the NCI Common Toxicity Criteria (CTCAE) version 3.0.
Time Frame: After 90 days post-treatment, up to 5 years per patient
Population: All enrolled patients that received SBRT therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT
Number analyzed (Participants) | 163
Participants | 0

3. Primary Outcome: Biochemical Disease-Free Survival Rate (bDFS)
Description: Biochemical Disease-Free Survival (bDFS) as defined by Phoenix and ASTRO. Biochemical progression-free survival events were defined as PSA of ≥ 0.4 ng/mL following postoperative radiotherapy, PSA > 2.0 ng/mL at any time, clinical progression, initiation of non-protocol hormone therapy, and death from any cause.
Time Frame: Up to 5 years
Population: All enrolled patients that received SBRT therapy with PSA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT
Number analyzed (Participants) | 163
Participants | 7

4. Secondary Outcome: Rate of Local Failure
Description: Proportion of patients with 'local failure', which is defined as clinical evidence local recurrence. Clinical failure includes a palpable abnormality that has increased in size, failure of regression of a palpable abnormality, or redevelopment of a prostate abnormality after complete response, further confirmed by prostate biopsy.
Time Frame: Up to 5 years
Population: Data were not collected.
Arm/Group | SBRT
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Distant Failure
Description: Proportion of patients with 'distant failure' (includes regional failure) which is defined as documented clinically via bone scan, CT or other imaging study that shows metastatic disease (disease located distant from the prostate area).
Time Frame: Up to 5 years
Population: Data were not collected.
Arm/Group | SBRT
Number analyzed (Participants) | 0

6. Secondary Outcome: 5-year Overall Survival (OS)
Description: Percentage of patients that remained alive 5 years after start of study treatment. Deaths were from any cause.
Time Frame: At 5 years
Population: All patients that received SBRT therapy.
Measure: Number; unit: percentage of participants
Arm/Group | SBRT
Number analyzed (Participants) | 163
percentage of participants | 93.87

7. Secondary Outcome: Quality of Life (QoL) - FACT-G - Prior to Therapy
Description: The Functional Assessment of Cancer Therapy- General (FACT-G) is a self-administered 27-item questionnaire designed to measure four domains of HRQOL in cancer patients. It is comprised of physical (PWB), social (SWB), emotional (EWB), and functional (FWB) well-being subscales: (PWB; 7-items, score range 0-28), (SWB; 7-items, score range 0-28), (EWB; 6-items, score range 0-24), (FWB; 7-items, score range 0-28). The FACT-G generates an overall score of 0-108). All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much) and asks information regarding the patients last 7 days.
Time Frame: Prior to start of therapy
Population: Patients that received SBRT therapy, that completed quality of life assessments Prior to therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT
Number analyzed (Participants) | 36
score on a scale
  PWB | 26.06019 (2.716213)
  SWB | 23.70186 (3.641432)
  EWB | 19.58 (4.449)
  FWB | 23.44 (5.417)
  FACTG | 92.78983 (12.323307)

8. Secondary Outcome: Quality of Life (QoL) - FACT-G - At 24 Months
Description: as for outcome 7
Time Frame: At 24 months (post-start of therapy)
Population: Patients that received SBRT therapy, that completed quality of life assessments Prior to therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT
Number analyzed (Participants) | 21
score on a scale
  PWB | 26.10 (2.791)
  SWB | 21.95238 (6.645819)
  EWB | 21.25 (3.370)
  FWB | 22.85 (5.824)
  FACTG | 93.15000 (14.605211)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of up to 5 years.
Arm/Group | SBRT
All-Cause Mortality (participants affected / at risk) | 15/163
Serious Adverse Events (participants affected / at risk) | 2/163
Other Adverse Events (participants affected / at risk) | 9/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=163)
Incontinence (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary frequncy (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT (N=163)
Diarrhea (Gastrointestinal disorders) | 5
Urinary frequency/urgency (Renal and urinary disorders) | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Other (Renal and urinary disorders) | 3
nocturia (Renal and urinary disorders) | 1
weak stream (Renal and urinary disorders) | 1
hypercholesteremia (Investigations) | 1
Burning - tip of penis (Skin and subcutaneous tissue disorders) | 1
anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT00977860/Prot_SAP_000.pdf